CLINICAL TRIAL: NCT05005468
Title: A Phase II Trial of Camrelizumab Combined With Famitinib for Adjuvant Treatment of Stage II-IIIA Non-small Cell Lung Cancer With High-risk for Relapse and no Driver Gene Mutation.
Brief Title: A Phase II Trial of Camrelizumab Combined With Famitinib for Adjuvant Treatment of Stage II-IIIA NSCLC.
Acronym: CAMFA-L
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Head of department, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-ADJ-IIT-SHR1210-FMTN
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: NSCLC
Keywords: NSCLC; II-IIIA
MeSH Terms: interventions — camrelizumab; famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab Combined With Famitinib (Experimental): Drug: Camrelizumab Drug: Famitinib
  Interventions: Drug: Camrelizumab; Drug: Famitinib
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is given on the first day of each cycle, intravenous drip.
  Other Names: SHR-1210
  Arms: Camrelizumab Combined With Famitinib
Drug: Famitinib — Famitinib is administered orally, once a day.
  Other Names: Famitinib Malate Capsules
  Arms: Camrelizumab Combined With Famitinib

SUMMARY:
This is a phase II, open-label, multi-cohort study, aiming to investigate safety and efficacy of Camrelizumab combined with famitinib for adjuvant treatment of stage II-IIIA non-small cell lung cancer with high-risk for relapse and no driver gene mutation.

DETAILED DESCRIPTION:
Immunotherapy has shown good efficacy in advanced NSCLC. The IMpower010 study has found that immune adjuvant therapy after postoperative chemotherapy can significantly prolong disease-free survival. A number of basic and clinical studies have found that anti-vascular drugs can improve the tumor immune microenvironment, and the combination of anti-vascular and immunotherapy may further improve the efficacy. In this study, postoperative NSCLC with a high risk of recurrence was screened out through ctDNA detection, and received Camrelizumab combined with famitinib or observation to observe the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, both male and female;
2. Standard surgical R0 resection and pathologically confirmed patients with stage II-IIIA (UICC/AJCC 7th edition lung cancer TNM staging) non-small cell lung cancer;
3. ECOG PS score 0-1 points;
4. EGFR, ALK gene wild type;
5. The function of major organs is normal, the following standards are met: a) Routine blood examination (under 14 days without blood transfusion and no hematopoietic stimulating factor drugs for correction): hemoglobin (Hb) ≥90g/L; absolute neutrophil count (ANC) ≥1.5×10^9/L; platelet (PLT) ≥100×10^9/L; white blood cell count (WBC) ≥3.0×10^9/L; b) Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN); serum total bilirubin (TBIL) ≤1.5×ULN; serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50ml/min; c) coagulation function: activated partial coagulation activity Enzyme time (APTT), international normalized ratio (INR), prothrombin time (PT)≤1.5×ULN; d) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥50%;
6. The estimated survival time is at least 1 year;
7. Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug; for men, it should be Surgical sterilization or consent to use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug;
8. The patient voluntarily participates and signs an informed consent form (or signed by a legal representative). It is expected to have good compliance and be able to cooperate with the research according to the requirements of the plan.

Exclusion Criteria:

1. Have received neoadjuvant chemotherapy, radiotherapy or adjuvant radiotherapy;
2. There is an unhealed wound or the risk of hemorrhage as judged by the investigator;
3. Even after drug treatment, hypertension is still poorly controlled (continuous increase in systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg);
4. Urine routine test indicates urine protein ≥(++), or 24-hour urine protein ≥1.0g;
5. Abnormal blood coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow preventive use of low-dose aspirin and low molecular heparin;
6. Patients at risk of gastrointestinal bleeding, including the following conditions: There are active peptic ulcer lesions and stool occult blood (++ ~ +++); Those who have a history of melena and hematemesis within 3 months; For fecal occult blood (+) or (+/-), it is necessary to review the stool routine within 1 week. Those who still (+) or (+/-) must undergo gastroscopy. If there is ulcer, bleeding disease, and The treating physician believes that there is a potential risk of bleeding;
7. Suffer from uncontrolled cardiac clinical symptoms or diseases, such as (1) NYHA II and above heart failure; (2) Unstable angina; (3) Myocardial infarction within 1 year; (4) Clinical significance Patients with supraventricular or ventricular arrhythmia requiring clinical intervention;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] test results are positive, HBV-DNA ≥ 500 IU/ml and abnormal liver function; hepatitis C is defined as hepatitis C antibody [HCV-Ab] positive, HCV-RNA higher than the detection limit of the analysis method and abnormal liver function) or combined hepatitis B and C co-infection ；
9. Suffer from any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (hormone replacement) Can be included after treatment)); patients with childhood asthma that have been completely relieved and do not require any intervention or vitiligo after adulthood can be included, but patients who require medical intervention with bronchodilators cannot be included;
10. Severe infection (such as intravenous infusion of antibiotics, antifungal or antiviral drugs required) within 2 weeks before the first administration, or unexplained fever >38.5°C during the screening period/before the first administration;
11. Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
12. Suffered from or accompanied with other systemic malignancies in the last 5 years, (except for cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer);
13. Have received a preventive vaccine or attenuated vaccine within 4 weeks before the first administration;
14. Those who are known to be allergic to any test drug or its excipients;
15. Pregnant and lactating patients, and reproductive patients are unwilling to take effective contraceptive measures;
16. Have a clear history of neurological or mental disorders, including epilepsy and dementia;
17. Patients who cannot swallow the study drug, such as chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis) and intestinal obstruction and other factors that affect drug intake and absorption;
18. Other circumstances deemed inappropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
DFS | 6-18 months
  Disease free survival

SECONDARY OUTCOMES:
OS | 30-48 months
  Overall survival
DFS at 2/3/5years | 2-5 years
  DFS at 2/3/5years

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No